CLINICAL TRIAL: NCT03673761
Title: Role of Myosteatosis in the Occurrence and Persistence of Residual Muscle Weakness in Patients With Acromegaly and Cushing's Syndrome. Study of the Mechanisms Involved
Brief Title: Muscle in Acromegaly and Cushing's Syndrome
Acronym: MAC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-MIO-2017-41
Record Dates: First submitted 2018-08-30; First posted 2018-09-17 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Cushing Syndrome; Acromegaly
Keywords: muscle weakness; myopathy
MeSH Terms: conditions — Cushing Syndrome; Acromegaly; Muscle Weakness; Muscular Diseases | interventions — Magnetic Resonance Spectroscopy; Absorptiometry, Photon; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cushing's syndrome: a) Patients with Sd Cushing (SC): 40 women (25-60 years) with SC, with controlled hypercortisolism after treatment and without clinical / biochemical signs of relapse for more than 5 years.
  This group will under go the following procedures:
  * muscle MRI
  * dual-energy x-ray absorptiometry
  * muscle ultrasounds
  * blood testing
  Interventions: Other: MRI, dual-energy, x-ray absorptiometry, muscle ultrasounds, blood testing
- acromegaly: b) Patients with acromegaly: 40 patients of both sexes (25-60 years) with GH / Insulin-like-Growth Factor (IGF-I) controlled after treatment and without clinical / biochemical signs of relapse for more than 5 years.
  This group will under go the following procedures:
  * muscle MRI
  * dual-energy x-ray absorptiometry
  * muscle ultrasounds
  * blood testing
  Interventions: Other: MRI, dual-energy, x-ray absorptiometry, muscle ultrasounds, blood testing
- Healthy controls: Controls: n = 40; normal healthy control paired by age, sex and BMI will be included.
  This group will under go the following procedures:
  * muscle MRI
  * dual-energy x-ray absorptiometry
  * muscle ultrasounds
  * blood testing
  Interventions: Other: MRI, dual-energy, x-ray absorptiometry, muscle ultrasounds, blood testing

INTERVENTIONS:
Other: MRI, dual-energy, x-ray absorptiometry, muscle ultrasounds, blood testing — 3.Dixon, T2 mapping MRI microRNAs

SUMMARY:
Cushing's syndrome (CS) and acromegaly determine myopathy and muscle weakness which persist long-term after control of hormone excess. Fatty infiltration in skeletal muscle (myosteatosis) is associated with muscle atrophy, frailty, and increased morbidity and mortality in several human models. The study is aimed at evaluating muscle structure in patients with controlled CS and acromegaly, and correlate it with functional tests of muscle strength. In addition, circulating molecules potentially mediating persistent myopathy in these patients will also be assessed.

DETAILED DESCRIPTION:
Prior chronic exposure to glucocorticoids or growth hormone (GH) determines fat infiltration and persistent impairment of muscle structure in "cured" patients with CS or acromegaly, respectively. All this leads to irreversible changes in muscle strength and performance, markedly affecting morbidity and quality of life of these patients. In particular, muscle weakness would contribute significantly to the development of severe arthropathy associated with excess GH, as well as deterioration of bone status and increased risk of fracture, as described in patients with either CS or acromegaly in remission. Our aim is to evaluate whether muscular MRI is a useful tool for the assessment of myopathy and myosteatosis in these patients. If this is the case, we would have identified a non-invasive test that would allow the follow-up of patients at risk of developing functional motor problems, anticipating the onset of muscle weakness or fatigue and consequent deterioration of their quality of life. On the other hand, we will examine the role of microRNAs, which can suppress the process of myogenic differentiation, as potential modulators of myopathy in these conditions. Indeed, microRNAs could be used in clinical practice as markers to identify patients at risk of myopathy, and develop strategies for their prevention. Clarifying the impact of muscle fat infiltration on muscle strength would allow us to better understand the interaction between muscle and adipose tissue, encouraging research on potential mediators of this relationship, such as myostatin (MSTN) (able to direct the mesenchymal cell muscle towards the formation of adipocytes at the expense of myocytes) and adiponectin (ApN) (which keeps the levels of fat in the muscle low while favoring the formation and regeneration of muscle tissue).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Cushing's syndrome or acromegaly who have been in remission for at least 5 years.

Exclusion Criteria:

* Pregnancy, breastfeeding, chronic liver/kidney disease, chronic treatment with glucocorticoids.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Patients with Sd Cushing (CS): 40 women (25-60 years) with CS, with controlled hypercortisolism after treatment and without clinical / biochemical signs of relapse for more than 5 years.
  2. Patients with acromegaly: 40 patients of both sexes (25-60 years) with GH / IGF-I controlled after treatment and without clinical / biochemical signs of relapse for more than 5 years.
  3. Controls: n = 60; normal healthy control paired by age, sex and BMI will be included.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
MRI assessment of fatty infiltration in tigh muscles. | Within one year since recruitment
  Quantitative muscle 3Tesla-MRI (mappting T2 and 3.Dixon) will be used. Assessment of fatty infiltration as well as measurement of necrosis and inflammation areas in tigh muscles will be performed.

SECONDARY OUTCOMES:
microRNAs | Within one year since recruitment
  A bioinformatic study will be carried out to select a set of miRNAs differentially expressed in acromegaly and Cushing's syndrome as compared with controls. The miRNAs will be selected according to the pathophysiological pathways (GO, KEGG) in which they are involved and taking into account the pathophysiology of Cushing's syndrome and acromegaly. Differentially expressed miRNAs will be then related to primary outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Please Select, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martel-Duguech L, Alonso-Jimenez A, Bascunana H, Diaz-Manera J, Llauger J, Nunez-Peralta C, Montesinos P, Webb SM, Valassi E. Prevalence of sarcopenia after remission of hypercortisolism and its impact on HRQoL. Clin Endocrinol (Oxf). 2021 Nov;95(5):735-743. doi: 10.1111/cen.14568. Epub 2021 Aug 6. PMID 34323296
- [Derived] Martel-Duguech L, Alonso-Jimenez A, Bascunana H, Diaz-Manera J, Llauger J, Nunez-Peralta C, Biagetti B, Montesinos P, Webb SM, Valassi E. Thigh Muscle Fat Infiltration Is Associated With Impaired Physical Performance Despite Remission in Cushing's Syndrome. J Clin Endocrinol Metab. 2020 May 1;105(5):dgz329. doi: 10.1210/clinem/dgz329. PMID 31912154